CLINICAL TRIAL: NCT00570999
Title: Randomised Placebo-Controlled Double-Blind Phase II Study Applying Palifermin to Improve T-cell Immune Reconstitution After Haploidentical Allogeneic Peripheral Blood Progenitor Cell (PBPC) Transplantation
Brief Title: Palifermin After Haploidentical PBSCT
Acronym: KGF Haplo Allo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Amgen (Industry)
Responsible Party: Kim Champion, EBMT (European Group for Blood and Marrow Transplantation)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCt: 2007-003241-32
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Non-Hodgkin's Lymphoma or Hodgkin's Disease; Acute Leukaemia; Myelodysplastic Syndrome; Chronic Myeloid Leukemia; Osteomyelofibrosis
Keywords: Peripheral blood stem cell transplantation; Palifermin; Kepivance; Prevenar; Placebo
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Fibroblast Growth Factor 7; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Palifermin once daily at a dose of 60 mg/kg/day for 3 days before the start of the conditioning regimen and then for 3 consecutive days starting on the day of transplantation (days 0 to day +2 inclusively).
  Interventions: Drug: Palifermin
- Arm B (Placebo Comparator): Placebo at a dose of 1.2 mL (saline 0,9%) once daily for 3 days before the start of the conditioning regimen and then for 3 consecutive days starting on the day of transplantation (days 0 to day +2 inclusively).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Palifermin — 60 mg/kg/day
  Other Names: Keratinocyte growth factor; Kepivacine
  Arms: Arm A
Other: Placebo — 1,2 mL once daily
  Other Names: 0.9% saline
  Arms: Arm B

SUMMARY:
This is a double blind, placebo controlled clinical trial, where patients with an advanced form of blood cancer are treated with haploidentical allogeneic peripheral blood progenitor cell (PBPC) transplant after which they are randomised to receive either placebo or a keratinocyte growth factor (Palifermin or Kepivance®).

The function of Kepivance® is to stimulate the growth of epithelial cells. This drug has also been suggested to have an ability to help improve the reconstitution, or development, of the immune system after the transplantation.

The hypothesis is that the patients T-cell dependent humoral immune response to recall antigen (PrevenarTM) will be higher in in palifermin treated patients than in the placebo control group

ELIGIBILITY:
Inclusion Criteria:

Recipient:

* Chemosensitive low/high grade B-NHL or T-NHL, Multiple Myeloma (MM) in partial or complete remission
* ALL and AML, secondary AML and biphenotypic acute leukemia in complete remission (CR1 or CR2) or PR (only if ≤20% blasts in BM), Myelodysplastic syndrome (MDS)
* CML in chronic or accelerated phase
* Osteomyelofibrosis (OMF)
* Hodgkin lymphoma (HD) in partial or complete remission
* Age ≥18 years, ≤ 65 years
* ECOG status ≤2
* Prior treatment with 3 or less different chemotherapy regimens (not cycles); prior local radiotherapy is allowed except radiation involving the thymus
* Adequate pulmonary function
* Left ventricular ejection fraction (LVEF) >30%
* Haploidentical related donor
* Failure to find matched related or matched unrelated donor and urgently requiring transplantation
* Planned conditioning regimen per Aversa or Würzburg protocol
* Women must be post-menopausal, sterile or use effective contraception and have a negative pregnancy test at study entry (β-HCG neg)
* Signed informed consent

Donor:

* Healthy family member
* Selection based on typing of HLA-A, B, C, DR loci. Donor must be at least genotypically HLA-A, B, C, DR haploidentical to the patient, but must differ for 2-3 HLA allele(s) on the unshared haplotype
* Donors must be capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central venous catheter should leukapheresis via peripheral vein be inadequate.
* Donors must agree to a 2nd donation of PBPCs in case of insufficient CD34+ cell collection or should patient fail to demonstrate sustained engraftment
* Signed informed consent

Exclusion Criteria:

Recipient:

* History of or concurrent cancer (< 5 years ago) other than those named in inclusion criteria
* Primary chemorefractory disease
* CML in blast crisis
* MM with no or minor response to previous treatment
* Prior treatment with palifermin, or other keratinocyte growth factors
* Documented hypersensitivity to palifermin, E. coli-derived proteins, or any component of the product
* Documented hypersensitivity to Prevenar vaccine or its components
* Prior allogeneic or tandem PBPC transplantation (no more than 1 previous autologous transplantation
* Prior total body irradiation
* Post thymectomy
* Major anticipated illness or organ failure incompatible with survival from PBPC transplantation
* Active chronic skin disease requiring therapy
* Active inflammatory bowel disease requiring therapy
* Active uncontrolled infection
* Sero-positive HIV
* Pregnancy or breast-feeding
* Active invasive fungal tissue infection (EORTC criteria)
* 30 days or less since receiving an investigational product or device in another clinical trial
* Concurrent enrolment in another trial is not permitted unless the purpose is for long-term follow-up/survival data only, or observational only
* Chronic pancreatitis or history of acute pancreatitis within 1 year prior to transplant
* Psychiatric disorder associated with incompliance
* Myocardial infarction less than 3 months pre enrolment or EF <30% as measured in echocardiography/laevoventriculography
* Infusion of retrovirally or other transduced cells are not permitted.
* Planned intravenous application of immunoglobulins is contraindicated throughout the study period.
* Donor lymphocyte infusions are not allowed.

Donor:

* A positive HIV or HTLV-1 test or evidence of active/persistent viral hepatitis infection.
* Evidence of any other active infection
* Any medical condition (i.e. insulin-dependent diabetes, cardiovascular disorders, chronic inflammatory diseases) posing a health risk for peripheral blood stem cell harvest
* Hematopoietic or marrow function related disease interfering with the collection of sufficient numbers of normal progenitor cells
* Pregnancy or breast-feeding
* Any malignancy besides basal cell epithelioma or cured malignancy < 5 years ago
* Psychiatric disorder associated with incompliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
To test palifermin's effect on the T-cell dependent humoral immune response to recall antigen (Prevenar™) | at study day +270 (20 days after the third Prevenar injection)

SECONDARY OUTCOMES:
To assess if Palifermin improves T-cell reconstitution after haploidentical allogeneic transplantation | at study days: +240
To assess if Palifermin improves T-cell reconstitution after haploidentical allogeneic transplantation | Study days +210, +240, +270
To assess disease free survival (DFS) and overall survival (OS), incidence and duration of GvHD, incidence and severity of OM, and incidence and severity of infections | at 2 years
To assess drug related safety | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Seggewiss, MD, Study Chair — University Hospital of Würzburg
Locations (1):
- Dr Ruth Seggewiss, Würzburg, Germany